CLINICAL TRIAL: NCT01641380
Title: Meaningful Use of Technology to Improve Health Care Delivery for Urban Adolescents: Focus on Teen Pregnancy Prevention (DepoText Study)
Brief Title: Meaningful Use of Technology to Improve Health Care Delivery
Acronym: DepoText
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Thomas Wilson Sanitarium for Children of Baltimore City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NA_00043284
Record Dates: First submitted 2012-07-10; First posted 2012-07-16 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-01

CONDITIONS: Contraceptive Behavior
Keywords: Depoprovera; Contraception; Appointment adherence/attendance; Pregnancy Prevention
MeSH Terms: conditions — Contraception Behavior | interventions — Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Adolescents in the Control Arm received standard of care. They continue to receive the DepoProvera injections through scheduled appointment, but would not receive a call from the nurse case manager regarding DepoProvera appointments until they have missed their scheduled DepoProvera appointment.
- Text Messaging Intervention (Experimental): Adolescents in the intervention arm receive text message reminders for appointments and positive sexual health messages regarding use of DepoProvera in between scheduled appointments. They are encouraged to seek care for assistance with obtaining condoms and/or if they are having problems with the medication.
  Interventions: Behavioral: Text Messaging Intervention

INTERVENTIONS:
Behavioral: Text Messaging Intervention — 1. Online enrollment in the Compliance for Life® (CFL) system through iReminder)
  2. Welcome Message 24 hrs after enrollment
  3. Appointment Reminder prior to 3 month injection cycles
  4. Monthly health reminders i. Condom use ii. Weight control iii. Side Effect Management 5.6-month STD testing reminder
  6.Call for missed appointment or no reply to appointment reminder (or other text message)
  Other Names: Compliance for Life®
  Arms: Text Messaging Intervention

SUMMARY:
While there have been major declines in teenage pregnancy around the country, Baltimore, Maryland has continued to experience increases over the last several years. Access and adherence to contraception has been found to be a major contributor to declines in teen pregnancy worldwide. The aim of this proof of concept pilot project is to determine preliminary efficacy of the DepoText Intervention. We will randomize urban adolescent girls who have elected Depo-Provera for ongoing contraception to receive either standard counseling and clinic appointment reminders or a text messaging (DepoTEXT) follow-up intervention. Participants in the DepoTEXT intervention will receive reminders for clinic visits and encouraging messages each month for STI prevention. The primary outcome is the preliminary efficacy for improving appointment adherence.

DETAILED DESCRIPTION:
Aims:

The aim of this proof of concept pilot project is to determine the feasibility and acceptability of a text messaging reminder system for communicating with urban adolescents using Depo-Provera for long-acting contraception. We will randomize urban adolescent girls who have elected Depo-Provera for ongoing contraception to receive either standard counseling and clinic appointment reminders or a text messaging (DepoTEXT) follow-up intervention. Participants in the DepoTEXT intervention will receive reminders for clinic visits and encouraging messages each month for STI prevention. The primary outcome is the preliminary efficacy for improving appointment adherence. Secondary measures include patient responsiveness to text messages and acceptability/satisfaction with this approach.

Setting and Participants:

This research study will be conducted in the Johns Hopkins Harriet Lane Clinic located Baltimore, Maryland. As noted above, Baltimore currently has rates of teen pregnancy that are significantly higher than statewide rates.5, 6 The United States Census estimates that there are 47,710 adolescents between the ages of 15-19 years in Baltimore. 7 Using 2007 Youth Risk Behavior Survey estimates, approximately 35,829 youth in this age group are having sexual intercourse and 13,302 are not using condoms for either STI or pregnancy prevention. 20 The current rise in birth rates to teens in urban Baltimore has prompted a joint initiative involving the mayor's office, Baltimore City Health Department, Urban Health Institute, and Healthy Teen Network.21

The Harriet Lane Clinic located in East Baltimore primarily serves low-income African American families from the neighboring communities. Adolescents and young adults in East Baltimore have high rates of pregnancy and STIs. During the 1st 12-months of funding of the Johns Hopkins Harriet Lane Teen Clinic's Title X Program, the majority of clients were females aged 15 to 25 years (83%), uninsured (52%), and minors seeking confidential services (50%). The program provides sexual/reproductive health services to young persons who are uninsured, underinsured and seeking confidential services. More than 80% of patients served by the clinic participate in a Medicaid Managed Care Organization. While there are approximately 250 individuals on the Depo-Provera logs, the Harriet Lane Clinic currently has more than 100 active users, but adherence to scheduled Depo-Provera appointments remains a problem despite access to care through our clinical site.

Recruitment:

Adolescent girls 13-21 who have 1) elected Depo-Provera for long-acting contraception and 2) have an active cell phone for their personal use will be asked by the adolescent nurse case manager and/or research staff at 1) routine clinical visits and 2) through telephone outreach if they would be willing to participate in a quality improvement intervention that involved random assignment to the text messaging intervention that reminds them of their next Depo-Provera visit via text message or the standard clinic reminders via phone.

All recruitment will take place in the confines of their private room during their routine clinical visits for family planning or via phone at the preferred contact number listed by the patient. The same degree of privacy will be afforded as during the clinical visit or during routine follow-up phone calls.

Randomization & Blinding As noted in the above schematic, adolescents who agree to participate will be randomized to the intervention or control arms at the time of enrollment. A computer-generated randomization sequence for block randomization (5 units) will be employed. Ordered envelopes will be generated for each enrollment packet to guide the research staff regarding group assignment.

Interventions All adolescents will receive care from the Harriet Lane Adolescent Medicine Clinic according to the existing clinical protocol. During "Depo visits" patients receive a nursing assessment, medical assessment if indicated, counseling, and if all is well their next injection, an appointment card with the date of the next injection. Patients are also offered automatic clinic reminders via their home phone. All adolescents in the study will complete a baseline interview and brief follow-up interview at each visit based on the standard interviews conducted by staff at each Depo-Provera visit. Adolescents who are enrolled by phone will be asked the questions via phone and then interviewed at the next visit.

In addition to standard of care and brief study interviews, adolescents in the Depo-TEXT intervention will be provided with online enrollment in the Compliance for Life® (CFL) system through iReminder) to receive a welcome Message 24 hrs after enrollment, appointment reminders prior to 3 month injection cycles, monthly health reminders (condom use, weight control on Depo-Provera, side effect management, 6-month STD testing reminder, call for text replies to reschedule missed appointments.) Intervention participants will receive standard of care for those enrolled in the Depo-Provera clinical program through which a nurse case manager responds to self-activated queries for assistance and missed clinic appointments.

Patients will be followed for adherence for 2-3 Depo-Provera injection cycles depending on the time of enrollment.

Human subjects Protections:

All participants will provide informed oral consent and/or via phone and will be informed that their participation in the study will have no effect on subsequent medical care. All patient data will be kept confidential and secure by using subject ID numbers, electronic collection of survey information and storage on secure servers with password protection for access. All research team members on this project have been educated in the protection of human research participants and the treatment of protected health information as evidenced by completion of their institutional compliance courses. Research assistants have completed the compliance courses as a part of their staff training. We are also using an established provider of global, secure and regulatory HIPAA compliant patient communication solutions to healthcare and biopharmaceutical research sectors to engage adolescents using SMS technology.

ELIGIBILITY:
Inclusion Criteria:

* Selected Depo-Provera for ongoing contraception
* Have a cell phone with text messaging capacity for personal use, and
* Agree to be randomized

Exclusion Criteria:

* Adolescent girls using other forms of contraception
* Adolescents who do not have a cell phone w/ text messaging capability for personal use

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Trent, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be made available to researchers for subsequent analyses. It will be available upon final completion of the study. Data can be obtained by submitting an initial query for review by the principal investigator.

REFERENCES:
- See also: Registration link on Johns Hopkins ICTR Trials Registry — http://trials.johnshopkins.edu/studyData.cfm?sdUUID=591B710E-D80A-1D0A-C128FF733488EB93

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research study was conducted in a large urban academic General Pediatric and Adolescent Medicine Practice in Baltimore, Maryland between October 2011 and February 2012.
Groups:
- Text Messaging Intervention: Adolescents in the intervention arm receive text message reminders for appointments and positive sexual health messages regarding use of DepoProvera in between scheduled appointments. They are encouraged to seek care for assistance with obtaining condoms and/or if they are having problems with the medication.
  Text Messaging Intervention:
  1. Online enrollment in the Compliance for Life® (CFL) system through iReminder)
  2. Welcome Message 24 hrs after enrollment
  3. Appointment Reminder prior to 3 month injection cycles
  4. Monthly health reminders i. Condom use ii. Weight control iii. Side Effect Management 5.6-month STD testing reminder
  6.Call for missed appointment or no reply to appointment reminder (or other text message)
Period: First Injection Cycle
Arm/Group | Control | Text Messaging Intervention
Started | 50 | 50
Completed | 43 | 44
Not Completed | 7 | 6
Period: Second Injection Cycle
Arm/Group | Control | Text Messaging Intervention
Started | 43 | 44
Completed | 39 | 38
Not Completed | 4 | 6
Period: Third Injection Cycle
Arm/Group | Control | Text Messaging Intervention
Started | 39 | 38
Completed | 36 | 33
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Youth assigned to the DepoText intervention arm also received a welcome text message, daily text appointment reminders using the Compliance for Life (CFL) ™ short messaging system (SMS) platform starting 72 hours before the clinical visit with the option to cease messages by responding (yes or no) with their plans to attend the visit. If the patient responded "no" to appointment reminders, then an email was automatically sent to the nurse case manager who contacted the patient to reschedule the appointment. Intervention adolescents also received prescheduled health messages regarding condom use for STI prevention, healthy weight management, encouragement to call the nurse for problems, and an STI screening reminder.
- Control: Standard of care
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 20 | 42
  Between 18 and 65 years | 28 | 30 | 58
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 48 | 50 | 98
  White | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Appointment Adherence (Efficacy)
Description: Participants who returned on-time for appointments
Time Frame: 9 months
Population: Evaluated differences in percentage of participants who return for on-time DepoProvera appointments for first cycle
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
participants | 34 | 28
Statistical Analysis 1: Comparison: Intervention vs Control; We also evaluated the difference between the number of days after the scheduled appointment patients returned; Test type: Superiority or Other; p < .05, Regression, Linear; Slope = -.75, 95% CI 2-sided [-1.4 to .06]
Statistical Analysis 2: Comparison: Intervention vs Control; On time for 1st follow-up visit; Test type: Superiority or Other; p = 0.5187, Chi-squared; Difference of proportions = 0.417, 95% CI 2-sided [-13.3307 to 24.8818] — Intervention 34/50; Control : 28/50

2. Primary Outcome: Responsiveness to Appointment Messages
Description: Overall responsiveness to delivery confirmation requests with A) Appointment messages and B) Informational Messages
Time Frame: 9 months
Population: Participants in the control group did not receive text messages (intervention) and so no data was collected for them.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 0
participants
  Responded to appointment messages | 38 |
  Responded to Informational messages | 34 |

3. Secondary Outcome: Proportion of Patients Satisfied With Messaging Service
Description: % of patients indicating satisfaction with the messaging reminder/health information service
Time Frame: 9 months
Population: Participants in the control group did not receive text messages (intervention) and so no data was collected for them.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 0
participants
  Satisfied with the program | 25 |
  Felt more connected to the clinic | 24 |

4. Other Pre Specified Outcome: Acceptability
Description: To determine acceptability we measured the number of individuals who were eligible for the trial and the number of eligible individuals who agreed to participate in the trial.
Time Frame: Baseline Recruitment
Population: Number of eligible participants among those approached
Measure: Number; unit: participants
Groups:
- Eligible Participants: Eligible participants among those approached for participation.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 116
participants | 100
Statistical Analysis 1: Comparison: Eligible Participants; Test type: Superiority or Other; [Proportion of Eligible Patients Enrolle = 0.948

ADVERSE EVENTS:
Arm/Group | Control | Text Messaging Intervention
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
1) Limited generalizability 2) Pilot study not powered to measure longitudinal efficacy; however, the preliminary data support expansion. 3) Data on duration of Depo- Provera use were not captured in enrollment data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes